CLINICAL TRIAL: NCT04027010
Title: A Randomized Controlled Trial of Virtual Student Health Center Among Incarcerated Juvenile Offenders
Brief Title: An Evaluation of Virtual Student Health Center Among Incarcerated Juvenile Offenders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WestEd (Other)
Collaborators: Oregon Youth Authority (Unknown); Efficacity (Unknown); The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8169
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Lack of Knowledge About Condoms and Birth Control; Adolescent Sexual Intercourse; Sexual Intercourse Without a Condom or Birth Control; Unplanned Pregnancies
Keywords: juvenile justice; male-focused intervention; unplanned teen fatherhood; technology-based intervention

STUDY DESIGN:
Intervention Model Description: The treatment condition involves participation in a teen pregnancy prevention program, Healthy U (formally known as Virtual Student Health Center). The comparison condition for the study is treatment as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Healthy U" tablet application (Experimental): Healthy U is a self-administered intervention implemented through a tablet app with interactive learning experiences, including videos, digital games, quizzes, and role-plays. Healthy U takes youth 3-4 hours to complete. The goals of Healthy U are to: 1) Increase male youth's perception of vulnerability to unplanned fatherhood, STDs and HIV; 2) Increase male youth's self-efficacy for negotiating condom use with their partners; 3) Increase male youth's self-efficacy for using condoms correctly and consistently every time they have sex; and 4) Increase male youth's engagement with goals and dreams for their future.
  Interventions: Other: "Healthy U" tablet application
- Treatment as usual (No Intervention): The counterfactual condition for the study is a business-as-usual condition. OYA does not provide much programming to youth in its facilities related to sexual health and pregnancy prevention.

INTERVENTIONS:
Other: "Healthy U" tablet application — There are seven modules in Healthy U: Puberty, Birth Control, Teen Pregnancy, HIV, STDs, Healthy Relationships, and Condom Negotiation. Each module has six sections: Introduction and Review, Narrative Teen Portrait, Information Film, Activity/Game, Dramatic Film, and Imagination Challenge. The Introduction and Review has videos lasting 1-2 minutes where the Healthy U "host" introduces each module. In the Narrative Teen Portrait for each module, a different teen discusses their experience with the topic for 1-3 minutes. The Information Film lasts 5-18 minutes per module and provides factual information. For each module, the Activity/Game includes multiple choice, true/false, or other games. The Dramatic Film lasts 5-17 minutes for each module and shows a fictional account of a teen experiencing the topic. Finally, the Imagination Challenge asks the youth to imagine a scenario, such as going to a health clinic to obtain free condoms.
  Other Names: Virtual Student Health Center
  Arms: "Healthy U" tablet application

SUMMARY:
WestEd and its partners Efficacity and the Oregon Youth Authority (OYA), are conducting a randomized controlled trial of an innovative teen pregnancy prevention program, Healthy U, for youthful male offenders. This study involves male teenagers (age 14-19) at high risk for involvement in risky sexual behavior, including teen pregnancy. The innovative, non-curricular, technology-based intervention, Healthy U, is self-directed, low-cost, user friendly, and offers great promise in reaching incarcerated youth. The purpose of this study is to test this intervention on a population of young men incarcerated at the OYA who will soon be released into the community. The intervention is tailored to this population by updating the design, videos, and examples to best reflect the youth in the study, and OYA staff are being trained to facilitate the self-guided intervention.

DETAILED DESCRIPTION:
WestEd and its partners, Efficacity and the Oregon Youth Authority (OYA), were funded by the Department of Health and Human Services (DHHS) to conduct a randomized controlled trial of an innovative teen pregnancy prevention program, Healthy U (formally known as Virtual Student Health Center), for youthful male offenders to test the impact of this innovative, non-curricular, technology-based intervention, that is self-directed, low-cost, user friendly, and offers great promise in reaching incarcerated youth. Healthy U was designed to give adolescents and teens the tools they need to reduce their risk of unintended pregnancy and sexually transmitted diseases (STDs), including HIV, using a low-cost, transportable platform that is user-friendly for youth (and staff to oversee). In this project, we take the innovative Healthy U intervention and modify its implementation for juveniles in custody of a correctional facility.

This study involved male teenagers (ages 14-19) at high risk for involvement in risky sexual behavior, including teen pregnancy. The findings from this study are intended to contribute to research on both teen pregnancy and crime prevention. Teen parents and their children are at greater risk for subsequent criminal offending, and the children of teen parents also have greater risk of child abuse and neglect victimization. The current knowledge base suggests that youth exposed to the juvenile justice system have sex more often with more partners at a younger age and without protection (Bryan, Rocheleau, Robbins, & Hutchinson, 2005). This randomized study was designed to contribute to our understanding of what works with this population and to strengthen our knowledge base around developing and implementing technology-based interventions in a juvenile correctional environment.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 14-19
* OYA commits
* Have the cognitive ability to complete the baseline and follow-up surveys
* Need to be within 30-90 days of release

Exclusion Criteria:

* Female
* Outside of age criteria
* Oregon Department of Corrections commits
* Does not have the cognitive ability to complete the baseline and follow-up surveys
* Not within 30-90 days of release

Ages: 14 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The study sample will include male youth who, at the time of recruitment, are incarcerated in one of the five OYA male juvenile justice facilities.
Enrollment: 295 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Sexual intercourse | 6 months after the baseline survey
  The outcome was based on four survey items. Youth who responded "no" to the first item: "Have you ever had sexual intercourse?" were coded as "0". Youth who responded "no" to the second item: "Have you been out of a close custody OYA facility any time in the past three months?" were also coded as "0". Youth who responded "no" to the third item: "During the last 3 months, did you have sexual intercourse, even once?" were also coded as "0". Youth who responded "yes" to the first three items and provided a valid response greater than zero to the fourth item: "In the last 3 months (include only the time you were outside of a close custody OYA facility), how many TIMES did you have sexual inter-course?" were coded as the value they entered.

SECONDARY OUTCOMES:
Sexual intercourse without a condom | 6 months after the baseline survey
  The outcome was created by subtracting the sexual intercourse outcome from the following measure based on four items. Youth who responded "no" to the first item: "Have you ever had sexual intercourse?" were coded as "0". Youth who responded "no" to the second item: "Have you been out of a close custody OYA facility any time in the past three months?" were also coded as "0". Youth who responded "no" to the third item: "During the last 3 months, did you have sexual intercourse, even once?" were also coded as "0". Youth who responded "yes" to the first three items and provided a valid response greater than zero to the fourth item: "In the last 3 months (include only the time you were outside of a close custody OYA facility), how many TIMES did you or your partner use a condom when you had sexual inter-course?" were coded as the value they entered. Youth who responded "none" to the fourth item were coded as "0".
Sexual intercourse without any methods of birth control | 6 months after the baseline survey
  The outcome was based on four survey items. Youth who responded "no" to the first item: "Have you ever had sexual intercourse?" were coded as "0". Youth who responded "no" to the second item: "Have you been out of a close custody OYA facility any time in the past three months?" were also coded as "0". Youth who responded "no" to the third item: "During the last 3 months, did you have sexual intercourse, even once?" were also coded as "0". Youth who responded "yes" to the first three items and provided a valid response greater than zero to the fourth item: "In the last 3 months (include only the time you were outside of a close custody OYA facility), how many times did you have sexual intercourse without you or your partner using any methods of birth control (that is, you didn't use a condom or any other type of birth control shown in the blue box above)?" were coded as the value they entered. Youth who responded "none" to the fourth item were coded as "0".
Subsequent pregnancies of female partners | 6 months after the baseline survey
  The outcome was created by subtracting the number of pregnancies reported at baseline from the number of pregnancies reported at the 6-month follow-up. At both time points, the measure was based on three questions. Youth who responded "no" to the first item: "Have you ever had sexual intercourse?" were coded as "0". Youth who responded "no" or "don't know" to the second item: "To the best of your knowledge, have you ever gotten someone pregnant, even if no child was born?" were also coded as "0". Youth who responded "yes" to the first two items and provided a valid response greater than zero to the third item: "To the best of your knowledge, how many times have you gotten someone pregnant?" were coded as the value they entered.

OTHER OUTCOMES:
Perceptions of condoms | 6 months after the baseline survey
  The outcome was calculated as the average response based on a scale of 1 (strongly disagree) to 5 (strongly agree) for the following four items:
  * Condoms should always be used if a person your age has sexual intercourse.
  * Condoms are a hassle to use.
  * Condoms are important to make sex safer.
  * Using condoms means you don't trust your sexual partner. Youth needed to complete three of the four items to be included in the calculation.
Perceptions of sexual intercourse | 6 months after the baseline survey
  The outcome was calculated as the average response based on a scale of 1 (strongly disagree) to 5 (strongly agree) for the following five items:
  * Having sexual intercourse is a good thing for you to do at your age. (Reverse coded)
  * At your age right now, having sexual intercourse would create problems.
  * At your age right now, not having sexual intercourse is important for you to be safe and healthy.
  * At your age right now, it is okay for you to have sexual inter-course if you use birth control, like a condom. (Reverse coded)
  * It is against your values to have sexual intercourse before marriage.
Confidence in use of birth control | 6 months after the baseline survey
  The outcome was the response on a scale of 1 (not at all confident) to 5 (completely confident) for the following item: "How confident are you that your partner used one of the methods of birth control shown in the blue box to the right the last time you had sexual intercourse?"
Intentions to use condoms | 6 months after the baseline survey
  The outcome was the response on a scale of 1 (no, definitely not) to 4 (yes, definitely) based on the following item: "If you were to have sexual intercourse in the next year, do you intend to use a condom?"
Intentions to use birth control | 6 months after the baseline survey
  The outcome was the response on a scale of 1 (no, definitely not) to 4 (yes, definitely) based on the following item: "If you were to have sexual intercourse in the next year, do you intend to have your partner use any of the methods of birth control shown in the blue box to the right?"
Knowledge about condoms | 6 months after the baseline survey
  The outcome was calculated as the average response based on a scale of 1 (not at all) to 3 (a lot) for the following three items:
  If a condom is used correctly, how much can it decrease the risk of…
  * Pregnancy?
  * Getting HIV, the virus that causes AIDS?
  * Getting chlamydia and gonorrhea? Responses of "don't know", which represented less than 6% of the data, were treated as missing. Youth needed to complete two of the three items to be included in the calculation.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - WestEd, Los Alamitos, California
  - WestEd, Woburn, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryan A, Rocheleau CA, Robbins RN, Hutchinson KE. Condom use among high-risk adolescents: testing the influence of alcohol use on the relationship of cognitive correlates of behavior. Health Psychol. 2005 Mar;24(2):133-42. doi: 10.1037/0278-6133.24.2.133. PMID 15755227